CLINICAL TRIAL: NCT04636931
Title: Morphological Changes of Plaque and Factors Influencing Plaque Healing After Drug-Coated Balloon for de Novo Coronary Lesions: A Optical Coherence Tomography Study
Brief Title: Serial Changes After Drug-Coated Balloon
Acronym: HEAL-aDCB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Principal Investigator, Da Yin, The director of the cardiology department, The First Affiliated Hospital of Dalian Medical University
Other Study IDs: HEAL-aDCB
Record Dates: First submitted 2020-10-16; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (5 ml) were collected before intervention using EDTA tubes at baseline and follow-up. Plasma samples were separated by centrifugation at 1000 g for 10 min and then stored at -80 °C until further analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims at evaluating the morphological changes of plaque estimated by optical coherence tomography (OCT) and Factors Influencing Plaque Healing after Drug-Coated Balloon (DCB) for de Novo Coronary Lesions.

DETAILED DESCRIPTION:
Percutaneous coronary intervention with a drug-eluting stent (DES) is the most common mode of revascularization for coronary artery disease. However, their efficacy is limited by in-stent restenosis and stent thrombosis. Drug-coated balloon (DCB) deliver an anti-proliferative drug into the vessel wall and leave nothing behind, which is a promising technique in the treatment of coronary artery disease. Previous many studies have confirmed that DCB treatment for de Novo coronary lesions is safe and efficient. But, data about morphological changes of plaque and factors influencing plaque healing after DCB for de Novo Coronary Lesions is scarce. The study compares morphological changes of plaques evaluated by OCT between baseline and 1-year follow-up and evaluates factors influencing plaque healing. All the included patient will receive dual antiplatelet therapy (DAPT) for one month followed by clopidogrel treatment.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosed as CAD underwent coronary angiography and OCT Examination.

* Patients with de novo lesion suitable for DCB treatment.
* The reference diameter of targeted artery ≥2.75mm, the length of targeted lesion ≤25mm.
* Agreed to accept DCB treatment and written the informed consent.

Exclusion Criteria:

* Patients with de novo lesion unsuitable for DCB treatment.
* In-stent restenosis, coronary dissection, coronary spam, thrombus
* left main artery disease
* Age>80 years old
* Cardiogenic shock or stroke admission
* Severe hepatic or renal dysfunction
* Poor quality of OCT image or massive thrombus
* Disagreed to accept DCB treatment.
* Life expectancy < 1year. Angiographic Exclusion Criteria
* After pre-dilation of targeted lesions, the patients with residual stenosis>30%, TIMI flow <III grade and presence of major dissection (C type or higher).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CAD patients
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Major cardiovascular adverse events rate | 1-year follow-up
  In patients treated by DCB, the safety objectives are to evaluate the occurrence of any adverse events in 1 year (re-infarction, re-hospitalization, revascularization by PCI or CABG, cardiac death, stoke, and major bleeding).

SECONDARY OUTCOMES:
Differences in lesion characteristics evaluated by OCT between baseline and follow-up. | 1-year follow-up
  Lesion characteristics evaluated by OCT include lipid-rich plaque, fibrous plaque, macrophage, cholesterol crystal, microchannels and calcification and minimal lumen area (MLA). The follow-up OCT assessment will be performed 12 months after the treatment procedure.
Differences in lipid-plaque characteristics evaluated by OCT between baseline and follow-up in setting of lipid-plaque. | 1-year follow-up
  The characteristics of lipid-plaque evaluated by OCT include lipid core length, mean lipid arc, max lipid arc, fibrous cap thickness (FCT). The follow-up OCT assessment will be performed 12 months after the treatment procedure.
The incidence of late lumen loss (LLL) at follow-up. | 1-year follow-up
  LLL is defined as MLA at follow-up - MLA at baseline < 0.
Differences in OCT-defined characteristics at baseline according to the presence of late lumen loss (LLL) at follow-up. | 1-year follow-up
  All the patients are divided into two groups according to presence of late lumen loss (LLL) at follow-up. The OCT-defined characteristics include plaque rupture, plaque erosion, lipid-rich plaque, fibrous plaque, macrophage, cholesterol crystal, microchannels and calcification. If the plaque is rich in lipid, the lipid core length, mean lipid arc, max lipid arc, fibrous cap thickness (FCT) will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: No